CLINICAL TRIAL: NCT02794818
Title: Penn State ProduceRx Feasibility Study: Developing a "Prescription Produce" Model That Can Impact Long-term Health Outcomes for Patients
Brief Title: Penn State ProduceRx Feasibility Study
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Sarayna Schock, MSII, Milton S. Hershey Medical Center
Other Study IDs: STUDY00005088
Record Dates: First submitted 2016-05-25; First posted 2016-06-09 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Dietary Modification
Keywords: Prevention; Nutrition

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Participating Patients: Participating patients will receive a prescription for weekly CSA produce boxes with nutritional education
  Interventions: Behavioral: Produce boxes with nutritional education
- Participating Providers: Participating providers will be surveyed at the end of the pilot to evaluate their perceived program efficacy, the benefit of the program to their patients, and elicit program feedback.

INTERVENTIONS:
Behavioral: Produce boxes with nutritional education — CSA produce boxes "prescribed" to study participants with free online nutritional education included
  Groups: Participating Patients

SUMMARY:
To provide "prescriptions" for weekly Community Supported Agriculture (CSA) boxes of fruits and vegetables to patients, accompanied by nutritional education (e.g. printed newsletters and YouTube videos), and evaluate benefits for participants by exploring commitment to the program, opinions about healthy eating, retention of nutrition and food preparation knowledge, overall takeaway from the program, as well as self-assessment of health status.

To establish the overall feasibility of an effective "prescription produce" program for at-risk and underserved patients - called "ProduceRx" - by utilizing produce from regional farms in addition to the resources of the Penn State Health System and an interdisciplinary team of healthcare workers (dietitians, dietetic interns, and medical students).

To provide a proof-of-concept for this model (i.e. ProduceRx + interdisciplinary approach to health education) for other healthcare institutions.

DETAILED DESCRIPTION:
Participating prescribers within the Penn State Health system will identify potential patients for ProduceRx based on the "high-risk" or "underserved" requirements. For the initial pilot starting on August 1, 2016, the following four physicians have agreed to participate with the program/study: Dr. Ann Rogers, Dr. Marsha Novick, Dr. Peter Lewis, and Dr. Laurie Nelson, whose specialties are general surgery and minimally invasive bariatric surgery, adolescent and bariatric medicine, family medicine, and internal medicine, respectively. Additionally, Lisa Hardy, a nurse practitioner at Dr. Ann Rogers' bariatric clinic, and Christine Bruce, a physician assistant at Dr. Laurie Nelson's internal medicine clinic will serve as the fifth and sixth prescribers. Prescribers will be provided with ProduceRx prescription pads that they will use to write "prescriptions" for their patients to the program. The prescription pads will be coded with a unique identifying code at the bottom that will allow researchers to keep track of data associated with that prescription (i.e. patient compliance with the program, difference in patient outcomes with different providers, etc.).

Patients will be recruited by the abovementioned physicians based on the physicians' interpretation of the two qualifications for the program: "high-risk" or "underserved." Recruiting materials such as informational brochures and advertisement signs (both electronic and printed) will be utilized to help these providers explain the program to qualifying patients without sacrificing time in the office. If selected patients elect to participate in the program, they will visit the ProduceRx website at https://sites.psu.edu/producerx and register for the program. Initial registration will feature an informed consent form to participate in research associated with this program. Patients will have the option of consenting or declining to consent to participation in this research. For those that consent, they will complete their initial survey through REDCap before bring routed to the participating farm's weekly ordering platform. Those patients who decline to consent will be automatically routed to the participating farm's ordering platform to order their first weekly box.

The survey will be a modified version of the CDC's Behavioral Risk Factor Surveillance System Questionnaire (BRFSS). This survey will assess patients' demographic characteristics, as well as health characteristics and behaviors. Demographic variables include age, race/ethnicity, education level, and employment status. Health characteristics include self-reported medical conditions, and height and weight (for calculation of body mass index). The survey will ask participants to self-report fruit and vegetable consumption and perceived barriers to consumption. Level of physical activity will also be monitored throughout the program to see if it is affected by changes in nutrition. Additionally, investigators will measure compliance of patients with the program; compliance will be defined as the number of weeks that patients voluntarily participate (purchase weekly boxes of produce) throughout the program from the time that they register with the program until the end of the pilot in December 2016.

During subsequent weeks, patients will visit the farm's website directly to order their weekly produce boxes. Participants will be asked to complete a post-program questionnaire at the end of the pilot in December 2016. Meanwhile, the main ProduceRx website will function as a platform for nutritional education delivery (delivered by medical students, registered dietitians, dietetic interns, as well as opportunities for other healthcare workers and community members), with links to the program's YouTube cooking/nutrition videos and postings of electronic versions of the printed newsletters. The website will also feature a calendar of upcoming local events, such as nature hikes, outdoor walks, free cooking classes, and farmers' markets, in order to facilitate an overall healthy lifestyle outside of the actual program. Additionally, the website will feature a comments section for participants to ask questions and communicate with one another. This comments section will be monitored to ensure appropriate commenting.

At the end of the program, a focus group will be held at Penn State Hershey Medical Center (PSHMC) to evaluate the functionality/feasibility of the pilot, including logistical convenience, how much produce was utilized each week, and what challenges participants faced integrating the produce and educational content into their daily lives. The focus group will ideally last from 45 to 90 minutes and will be moderated by Sarayna Schock, an MSII and PI on this study. A semi-structured interview guide will be used and responses will be recorded to adequately capture all feedback. These focus group responses will be recorded and transcribed by research volunteers and analyzed by an interdisciplinary research team to identify emergent themes.

To ease the burden of time constraints already imposed on physicians, participating healthcare providers will be surveyed via email at the end of the pilot to evaluate their perceived program efficacy, the benefit of the program to their patients, and elicit program feedback. A semi-structured survey created with REDCap will be used to solicit specific responses, in addition to open feedback.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals (ages 18-75) who are currently patients in the Penn State Hershey Health system in the departments of Family and Community Medicine, General Pediatrics, Internal Medicine, General Surgery and Minimally Invasive Surgery/Bariatric, Endocrinology, and Cardiology.
2. Individuals at risk for developing chronic illness and metabolic disease as identified by PCP, care coordinator, or a participating physician from an abovementioned specialty.
3. Individuals willing to participate in the program and complete a pre-program survey and a post-program survey in December 2016.
4. Individuals with access to transportation to and from the CSA drop-off sites.
5. Individuals willing/able to pay the $10 subsidized "copay" for the weekly box of produce (federal food stamps in the form of SNAP/EBT vouchers will be accepted by Strites Orchard as a means of payment).
6. Individuals that speak English.
7. Individuals with difficulty obtaining fresh produce or lack of knowledge regarding healthy cooking methods and nutrition, as determined by PCP or a participating physician from an abovementioned specialty.
8. Prescribers (physicians, nurse practitioners, and physician assistants) in the Penn State Hershey Health system in the departments of Family and Community Medicine, General Pediatrics, Internal Medicine, General Surgery and Minimally Invasive Surgery/Bariatric, Endocrinology, and Cardiology.

Exclusion Criteria:

1. Individuals outside of immediate areas of Strites Orchard's CSA drop-off sites (which include the following: Bosler Avenue, Lemoyne; Koch Lane Harrisburg (Paxtonia); Allendale, Camp Hill; Strites Orchard, Harrisburg; Dogwood Lane, Dillsburg; East Willow Street, Elizabethtown; Hampden Summit; Linglestown Rd., Harrisburg; St. Johns Drive, Camp Hill; Shetland Dr., Hummelstown; West Areba Ave., Hershey; Wickerberry Lane, Palmyra; W. Green St., Mechanicsburg; Brisban St. Harrisburg (Paxtang); Cattell St., Middletown; and N. 2nd St., Harrisburg.)
2. Individuals unaffiliated with the Penn State Hershey Health System.
3. Individuals who already have sufficient fruits and vegetables in their diet as determined by the participating physician.
4. Non-English speaking participants.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients determined to be "underserved" or "at-risk" within the Penn State Health System
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Modified CDC BRFSS Survey | 18-week study period
  Questionnaire items will assess participants' demographic characteristics, health characteristics, and behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Milton Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kraschnewski JL, George DR, Rovniak LS, Monroe DL, Fiordalis E, Bates E. Characterizing customers at medical center farmers' markets. J Community Health. 2014 Aug;39(4):727-31. doi: 10.1007/s10900-014-9818-x. PMID 24421001
- See also: Main ProduceRx program website — https://sites.psu.edu/producerx